CLINICAL TRIAL: NCT00931437
Title: Absorption of Different Forms of Vitamin K From Dairy Products
Brief Title: Vitamin K-absorption From Dairy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Dr. C. Vermeer, VitaK BV
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-3-086
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: vitamin K; Bio-availability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vitamin K-rich dairy product (Experimental): one single intake of a dairy product containing several K-vitamins: phylloquinone, menaquinone-7,8,9-and 10.
  Interventions: Dietary Supplement: vitamin K-rich dairy product

INTERVENTIONS:
Dietary Supplement: vitamin K-rich dairy product — several forms of vitamin K: phylloquinone, menaquinone-7,-8,-9,and -10.

SUMMARY:
Lactic acid bacteria produce a mixture of higher menaquinones, including menaquinone-9 (MK-9) and menaquinone-10 (MK-10). Vitamin K1 (phylloquinone) is normally present in chloroplasts in green vegetables. A new dairy product is developed containing both vitamin K1 and K2-vitamins. However, the extent to which the various forms of vitamin K are absorbed from such a mixture is not known. In this study the absorption profile of phylloquinone and menaquinones from this new dairy product containing several K-vitamins is investigated. This study describes a dietary intervention experiment for one single cocktail containing several K-vitamins as part of a dairy product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 20 and 45 years old
* Subjects of normal body weight and height according to BMI < 30
* Subjects of Caucasian race
* Subject has given written consent to take part in the study

Exclusion Criteria:

* Subjects with (a history of) metabolic or gastrointestinal disease
* Subjects presenting chronic degenerative and/or inflammatory disease
* Abuse of drugs and/or alcohol
* Subjects receiving corticoid treatment
* Subjects using oral anticoagulants

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
serum vitamin K levels: phylloquinone, menaquinone-7,-8,-9,and -10 | one single intake

SECONDARY OUTCOMES:
distribution of vitamin K-forms over lipoprotein fractions: triglyceride rich lipoprotein (TGRLP), intermediate-density lipoprotein (IDL), low-density lipoprotein (LDL), high density lipoprotein (HDL) as well as the lipoprotein-free fraction (LPF) | one single intake

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — VitaK / University of Maastricht
Locations (1):
- VitaK BV / University of Maastricht, Maastricht, Netherlands